CLINICAL TRIAL: NCT00274547
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Trial Assessing the Proportion of Patients Experiencing an Exacerbation and Proportion of Patients Hospitalized for an Exacerbation Over 6 Months During Treatment With Tiotropium 18 Mcg Capsule Once Daily in Patients With COPD in a Veterans Affairs Setting
Brief Title: Tiotropium (18 Mcg) Once Daily Via the HandiHaler® in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.266
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
The primary objective of this trial is to determine whether treatment with tiotropium (18 mcg) capsule once daily via the HandiHaler reduces the proportion of patients with COPD experiencing an exacerbation and the proportion of patients hospitalized for an exacerbation during a six month observation period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1829 (Actual)
Dates: Start 2001-09; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients experiencing an exacerbation | 6 months
Percentage of patients hospitalized for a COPD exacerbation | 6 months

SECONDARY OUTCOMES:
Time to first COPD exacerbation | 6 months
Time to first hospitalization associated with an COPD exacerbation | 6 months
Total number of days of corticosteroids for an COPD exacerbation | 6 months
Total number of antibiotics for an COPD exacerbation | 6 months
Number of unscheduled out-patient visits | 6 months
Total number of hospital admissions and total hospital days | 6 months
Trough post-dose FEV1 and FVC | after 3 and 6 months
90 minute post-dose FEV1 and FVC | after 3 and 6 months
Occurrence of serious adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (26):
- United States (26):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tuscon, Arizona
  - VA Long Beach Healthcare System, Long Beach, California
  - Boehringer Ingelheim Investigational Site, Palo Alto, California
  - Respiratory Diseases (111A), Bay Pines, Florida
  - J. Hillis Miller Health Center, Gainesville, Florida
  - Veteran Affairs Medical Center, Hines, Illinois
  - Veterans Affairs Medical Center, North Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 4720 I-10 Service Road, Metairie, Louisiana
  - Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - Veteran Affairs Medical Center, Minneapolis, Minnesota
  - Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - Boehringer Ingelheim Investigational Site, Reno, Nevada
  - Boehringer Ingelheim Investigational Site, Buffalo, New York
  - Bronx VA Medical Center, New York, New York
  - Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - Dallas VAMC, Dallas, Texas
  - Veterans Affairs Medical Center, Houston, Texas
  - Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - Hampton VA Medical Center, Hampton, Virginia
  - Hunter Holmes McGuire Medical Center, Richmond, Virginia